CLINICAL TRIAL: NCT02604797
Title: Analgesia Effects of Nalbuphine vs Sulfentanil in Patient-controlled Intravenous Analgesia After Cesarean Section
Brief Title: Analgesia Effects of Nalbuphine vs Sulfentanil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Sun Shen, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SShen
Record Dates: First submitted 2015-10-26; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: C.Delivery; Surgery (Previous), Gynecological
MeSH Terms: interventions — Nalbuphine; Sufentanil; flurbiprofen axetil; ramosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nalbuphine (Experimental): Nalbuphine group: nalbuphine 100 mg, ramosetron 0.3mg, background dose 1ml/h,patient-controlled analgesia(PCA) 1ml/time, lockout time 10 min, flurbiprofen axetil 50mg 6h after operation.
  Interventions: Drug: Nalbuphine; Drug: flurbiprofen axetil; Drug: ramosetron
- Sufentanil (Experimental): Sufentanil group: sufentanil 100ug, ramosetron 0.3mg, background dose 1ml/h, PCA 1ml/time, lockout time 10 min, flurbiprofen axetil 50mg 6h after operation.
  Interventions: Drug: Sufentanil; Drug: flurbiprofen axetil; Drug: ramosetron

INTERVENTIONS:
Drug: Nalbuphine — patient-controlled intravenous analgesia
  Other Names: nalbuphine 100 mg
  Arms: Nalbuphine
Drug: Sufentanil — patient-controlled intravenous analgesia
  Other Names: sufentanil 100ug
  Arms: Sufentanil
Drug: flurbiprofen axetil — patient-controlled intravenous analgesia
  Other Names: flurbiprofen axetil 50mg
Drug: ramosetron — patient-controlled intravenous analgesia
  Other Names: ramosetron 0.3mg

SUMMARY:
Cesarean section may result in great trauma and postoperative pain. Besides incision pain, uterine contraction pain is another source of postoperative pain after cesarean section. In clinical practice, a large amount of uterine contraction agent is routinely applied after cesarean section so as to promote involution of uterus and reduce postoperative hemorrhage, which also causes great uterine contraction pain. Acute pain is the risk factor of chronic pain, and may postpone the recovery from labour and influence the quality of life of parturient. Though various analgesia modules have been attempted, more than 20% parturients still experience severe postoperative pain, and pain management after cesarean section remains a challenge to anesthesiologists.

This study aim to compare the effects of nalbuphine hydrochloride vs sufentanil citrate on patient-controlled intravenous analgesia after cesarean section.

DETAILED DESCRIPTION:
Cesarean section may result in great trauma and postoperative pain. Besides incision pain, uterine contraction pain is another source of postoperative pain after cesarean section. In clinical practice, a large amount of uterine contraction agent is routinely applied after cesarean section so as to promote involution of uterus and reduce postoperative hemorrhage, which also causes great uterine contraction pain. Acute pain is the risk factor of chronic pain, and may postpone the recovery from labour and influence the quality of life of parturient. Though various analgesia modules have been attempted, more than 20% parturients still experience severe postoperative pain, and pain management after cesarean section remains a challenge to anesthesiologists.

Opiate drugs constitute the baseline medication for postoperative analgesia. However, pure μ opioid receptor agonist like morphine and fentanyl may induce adverse effects such as nausea, vomiting, dizziness, drowsiness and respiratory depression. Nalbuphine hydrochloride is an opiate-like substance structure-related oxymorphone, which is a κ receptor agonist/μ receptor partial antagonistic type analgesia drug. Specific κ receptor agonist and gene knockout experiment reveals that κ receptor agonist depresses the visceral pain induced by chemical stimulation, the effect of which outperforms pure μ opioid receptor agonist. Studies have discovered that some κ receptor agonists can reduce or inhibit the side effects of μ receptor agonist such as tolerance or dependence. The adverse effects of μ receptor agonist such as pruritus, nausea, vomiting, delayed gastric emptying are caused by the drug on peripheral opioid receptor, and can be relieved by opioid receptor agonist. The structure of nalbuphine hydrochloride is related to naloxone, an opioid receptor antagonist, therefore, the incidence of adverse effects of nalbuphine hydrochloride is lower than that of μ receptor agonist. In recent years, nalbuphine hydrochloride has become more and more popular in postoperative analgesia. There has been reports on intrathecal administration of nalbuphine hydrochloride for analgesia after cesarean section, while the effect of intravenous administration of nalbuphine hydrochloride on analgesia after cesarean section remains undetermined. This study aim to compare the effects of nalbuphine hydrochloride vs sufentanil citrate on patient-controlled intravenous analgesia after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* For primipara with selective cesarean section

Exclusion Criteria:

* Severe preeclampsia,
* pregnancy complicated with diabetes mellitus
* pregnancy complicated with cardiac disease,
* gestation age<37W
* recently use of opiate drugs or nonsteroidal antiinflammatory drugs within 48 h before operation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores of nalbuphine group | up to 24 months
Pain scores of sufentanil group | up to 24 months

SECONDARY OUTCOMES:
Usage of nalbuphine of nalbuphine group | up to 24 months
Usage of sufentanil of sufentanil group | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, Study Director — Department of Anesthesiology, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China